CLINICAL TRIAL: NCT06758596
Title: Research Investigating Drug Effects-2 (RiDE-2)
Acronym: RiDE-2
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY2024-0596
Record Dates: First submitted 2024-12-26; First posted 2025-01-06 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cannabis Use; Substance Use Disorder (SUD); Healthy
MeSH Terms: conditions — Substance-Related Disorders | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo oral capsule (Placebo Comparator): Participants will receive a placebo at their first or second laboratory visit.
  Interventions: Drug: Placebo Oral Capsule
- THC (Experimental): Participants will receive THC (7.5 mg) at their first or second laboratory visit.
  Interventions: Drug: THC

INTERVENTIONS:
Drug: Placebo Oral Capsule — A capsule that contains only dextrose filler administered during the first or second laboratory visit.
  Arms: Placebo oral capsule
Drug: THC — A capsule that contains 7.5 mg of THC as well as dextrose filler administered during the first or second laboratory visit.
  Arms: THC

SUMMARY:
The purpose of this study is to better understand how people's mood, behavior, and brains respond to different recreational drugs. We are also trying to understand why some people may feel differently or their brain may respond differently than other people after taking the same recreational drug.

ELIGIBILITY:
Inclusion Criteria:

* age 18-21 at eligibility visit
* body mass index of 18.5-30
* report using cannabis ≥10 times in their life and ≥1 time in the past 3 months, but <7 days a week (daily)
* medically and neurologically healthy
* score of ≥0.25 on the Personality Inventory for DSM-5 (PID-5) Anhedonia subscale

Exclusion Criteria:

* positive urine drug screen (UDS; except for THC) and/or positive saliva THC test
* contraindication for fMRI BOLD study (e.g., metal implants)
* severe mental illness (e.g., psychosis, mania, lifetime moderate-to-severe SUD (including moderate-to-severe CUD))
* heavy nicotine use in the past month (>20 cigarettes per week or electronic nicotine delivery system (ENDS) use equivalent
* night shift work
* females who are currently pregnant confirmed by urine pregnancy test, are planning pregnancy, or are lactating
* unwilling/unable to sign informed consent document
* current or past allergic or adverse reaction or known sensitivity to cannabinoid-like substances (Dronabinol/Marijuana/Cannabis/THC, cannabinoid oil, sesame oil, gelatin, glycerin, and titanium dioxide)
* physical or neurological diagnoses (e.g., cancer, diabetes, seizure disorder, Parkinson's, Multiple Sclerosis, loss of consciousness >10 min., etc.) that in the opinion of the Study Physician and Investigators could increase safety risks or influence the findings
* currently taking any medication that could interact with a single dose of Δ9-THC

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-07-15 (Estimated); Primary Completion 2031-03 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Recent Substance Use | Baseline screening, baseline drug administration, and every 6 months over two years of follow-up
  Participants will complete the 6-month Timeline Follow-Back (TLFB) and Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis Use Inventory (DFAQ-CU) to assess recent substance use. This measure will capture the frequency of substance use during the past 6 months, with greater values indicating more frequent substance use.
CUD/SUD Symptoms | Baseline screening and yearly over the two-year follow-up.
  Participants will complete the SCID CUD diagnosis and symptom assessment at baseline screening and yearly follow-ups to evaluate the presence and severity of cannabis use disorder (CUD) and other substance use disorder (SUD) symptoms.
Neural Reward Anticipation - fMRI response to reward anticipation (MID) | First and second laboratory visits, around 90 minutes to 2 hours after drug administration.
  Participants will complete the Monetary Incentive Delay (MID) task during fMRI scanning to assess neural activation related to reward anticipation. Greater activation in reward-related brain regions (e.g., striatum, prefrontal cortex) indicates greater neural sensitivity to anticipated rewards and the impact of THC on reward processing.
Computationally-Derived Behavioral Reward Learning Rate - Learning rate (alpha parameter) | First and second laboratory visits, around 90 minutes to 2 hours after drug administration.
  Participants will complete the Bandit task during fMRI scanning. A behavioral measure of learning rate (alpha parameter) will be derived from computational models based on the Rescorla-Wagner (RW) model, with higher learning rates indicating greater learning and adaptation to reward contingencies.
Computationally-Derived Behavioral Reward Sensitivity - Reward sensitivity (inverse temperature parameter) | First and second laboratory visits, around 90 minutes to 2 hours after drug administration.
  Participants will complete the Bandit task during fMRI scanning, and a behavioral measure of reward sensitivity will be derived from the Rescorla-Wagner (RW) model. Greater values indicate higher sensitivity to rewards and a stronger preference for rewarding outcomes.
Neural Encoding of Reward Prediction Errors - fMRI response to reward prediction errors (Bandit Task) | First and second laboratory visits, around 90 minutes to 2 hours after drug administration.
  Participants will complete the Bandit task during fMRI scanning. fMRI analysis will focus on trial-wise neural encoding of prediction errors, with greater activation indicating more salient reward learning signals in response to prediction errors, reflecting how the brain processes unexpected outcomes during reward learning.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic, clinical, behavioral, and fMRI data will be collected from 144 adults. All data will be de-identified prior to receipt by the repository, but the information needed to generate a global unique identifier (GUID) for the NIMH Data Archive (NDA) will be collected for each participant.
Supporting Information: Study Protocol, CSR
Time Frame: All data will be deposited to NDA starting 12 months after study begins and will be deposited every six months thereafter following the usual NDA data submission dates until the end of the study.
Access Criteria: To request access of the data, researchers will use the standard processes at NDA, and the NDA Data Access Committee will decide which requests to grant. The standard NDA data access process allows access for one year and is renewable.
URL: https://nda.nih.gov